CLINICAL TRIAL: NCT05315622
Title: Effects of the T12-L1 Vertebral Manipulation on Body Temperature, Arterial Tension and Cardiac Frequency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Collaborators: UCAM university (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLM012022
Record Dates: First submitted 2022-03-17; First posted 2022-04-07 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-03

CONDITIONS: Healthy Subjects; Spinal Manipulation; Manual Therapy

STUDY DESIGN:
Intervention Model Description: Single-blinded Randomized Controlled Trial
Who Masked: Participant
Masking Description: Participants will be unaware of their group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Bilateral vertebral manipulation of the T12-L1 vertebra
  Interventions: Other: Bilateral vertebral manipulation of the T12-L1 vertebra through manual therapy
- Placebo (Placebo Comparator): Application of slight manual tension to the vertebra without reaching a manipulation thrust
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Bilateral vertebral manipulation of the T12-L1 vertebra through manual therapy — Bilateral vertebral manipulation of the T12-L1 vertebra through manual therapy
  Arms: Intervention
Other: Placebo — Manual tension without reaching the manipulation "thrust"
  Arms: Placebo

SUMMARY:
Single-blinded Randomized Controlled Trial conducted amongst a sample of healthy subjects divided into two different groups: the experimental treatment will consist in bilateral T12-L1 vertebral manipulation, whereas the control group will receive a sham intervention consisting solely in applying tension without properly manipulating. Body temperature, arterial tension and cardiac frequency will be measured before and after the intervention. Changes in the aforementioned variables will be measured.

DETAILED DESCRIPTION:
The current study will correspond to a single-blinded Randomized Controlled Trial with two arms, conducted amongst a sample of healthy subjects, who will be divided into two different groups: the experimental treatment will consist in bilateral T12-L1 vertebral manipulation, whereas the control group will receive a sham intervention consisting solely in applying tension without properly manipulating. Three different variables will be measured prior to and after the intervention: body temperature, arterial tension and cardiac frequency, to subsequently calculate possible changes in the variables, with the aim of establishing the effect of the manipulation and/or sham treatment.

ELIGIBILITY:
Inclusion Criteria:

* Both genders;
* Over 18 years of age;
* Minimal amount of exercise per week: 1 hour/week;
* Covid-related aspects: Negative antigen-test 24 hours before the test or negative PCR 48 hours before the test.

Exclusion Criteria:

* Surgical intervention in the 5 years previous to the study;
* Any acute or chronic medical condition;
* Any pharmacological treatment;
* Osteosynthetic implants.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Body temperature | Change from baseline Body Temperature to ten minutes after the intervention
  Body temperature: Celsius degree will be measured by means of a digital thermometer
Body temperature | Change from baseline Body Temperature to seven days after the intervention
  Body temperature: Celsius degree will be measured by means of a digital thermometer
Cardiac frequency | Change from baseline Cardiac Frequency to ten minutes after the intervention
  Cardiac frequency: Beats per minute will be measured by means of OMRON M4 device, in compliance with the European Directive 93/42/EEC
Cardiac frequency | Change from baseline Cardiac Frequency to seven days after the intervention
  Cardiac frequency: Beats per minute will be measured by means of OMRON M4 device, in compliance with the European Directive 93/42/EEC
Arterial tension | Change from baseline arterial tension to ten minutes after the intervention
  Arterial tension (systolic/diastolic) will be measured by means of OMRON M4 device, in compliance with the European Directive 93/42/EEC
Arterial tension | Change from baseline arterial tension to seven days after the intervention
  Arterial tension (systolic/diastolic) will be measured by means of OMRON M4 device, in compliance with the European Directive 93/42/EEC

CONTACTS AND LOCATIONS:
Locations (1):
- UCAM, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be available to other researchers